CLINICAL TRIAL: NCT06957366
Title: Perioperative Anticoagulant Use for Surgery Evaluation -2 (PAUSE-2) Study Patients Receiving a Direct Oral Anticoagulant (DOACs-Dabigatran, Rivaroxaban, Apixaban or Edoxaban) and Needing Elective High-Bleed-Risk Surgery or an Invasive Procedure: A Randomized Control Trial
Brief Title: Perioperative Anticoagulant Use for Surgery Evaluation -2 (PAUSE-2) Study Patients Receiving a Direct Oral Anticoagulant (DOACs-Dabigatran, Rivaroxaban, Apixaban or Edoxaban) and Needing Elective High-Bleed-Risk Surgery or an Invasive Procedure
Acronym: PAUSE 2 RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, James Douketis, Dr. James Douketis-Principal Investigator, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAUSE 2 RCT (CTO 4938)
Record Dates: First submitted 2025-04-25; First posted 2025-05-04 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Atrial Fibrillation (AF); VTE
Keywords: anticoagulation; atrial Fibrillation; Surgery; Oral Anticoagulant; Blood thinner; DOAC; VTE; Interruption; PAUSE
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Patients taking Apixaban, Dabigatran, Rivaroxaban or Edoxaban will be randomly assigned to follow 1) PAUSE or 2) ASRA perioperative DOAC management.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Apixaban (Active Comparator): Patients currently taking Apixaban that have atrial fibrillation or Venous Thromboembolism and require an elective high bleed risk surgery or neuraxial anesthesia.
  Interventions: Other: PAUSE Perioperative DOAC Management; Other: ASRA Perioperative DOAC Management
- Dabigatran (Active Comparator): Patients currently taking Dabigatran that have atrial fibrillation or Venous Thromboembolism and require an elective high bleed risk surgery or neuraxial anesthesia.
  Interventions: Other: PAUSE Perioperative DOAC Management; Other: ASRA Perioperative DOAC Management
- Rivaroxaban (Active Comparator): Patients currently taking Rivaroxaban that have atrial fibrillation or Venous Thromboembolism and require an elective high bleed risk surgery or neuraxial anesthesia.
  Interventions: Other: PAUSE Perioperative DOAC Management; Other: ASRA Perioperative DOAC Management
- Edoxaban (Active Comparator): Patients currently taking Edoxaban that have atrial fibrillation or Venous Thromboembolism and require an elective high bleed risk surgery or neuraxial anesthesia.
  Interventions: Other: PAUSE Perioperative DOAC Management; Other: ASRA Perioperative DOAC Management

INTERVENTIONS:
Other: PAUSE Perioperative DOAC Management — PAUSE management is simple and easy to apply as patients having a high-bleed-risk surgery/neuraxial procedure interrupt DOACs for 2 days before and 2 days after surgery without heparin bridging or DOAC level testing.
Other: ASRA Perioperative DOAC Management — ASRA management is more complex, requiring 72-120 hours DOAC interruption and, in selected patients, pre-operative heparin bridging and DOAC level testing.

SUMMARY:
PAUSE 2 study is a prospective, open-label, blinded-endpoint non-inferiority RCT of PAUSE vs. ASRA management in DOAC treated high risk patients with AF/VTE who need elective high bleed risk surgery/procedure and/or any procedure involving neuraxial anesthesia. The purpose of the PAUSE 2 study is to show that PAUSE management will be as safe (i.e., non-inferior) as ASRA management, with 95% of patients having low/undetectable pre-operative DOAC levels <30 ng/mL in each group., at the time of surgery/neuraxial.

DETAILED DESCRIPTION:
As use of direct oral anticoagulants (DOACs) continues to increase so too will the need to manage such patients who require a surgery/procedure. Perioperative DOAC management is established and guideline supported in patients who need a low/moderate-bleed-risk surgery/procedure (e.g., hernia repair, colonoscopy), but there is uncertainty about managing high-risk patients who need a high-bleed-risk surgery (e.g., orthopedic, cardiac) or any neuraxial (i.e., spinal, epidural) anesthesia/procedure. The management of patients who are taking a DOAC (apixaban, dabigatran, edoxaban, rivaroxaban) and need a surgery/procedure is common, and will increase due to an ageing population and an associated increase in DOAC use. PAUSE-2 is applicable to approximately 96K patients/year in Canada, based on 1.6M prevalent patients with AF or VTE, of whom approximately 90% are taking a DOAC. Of these about 20% (approximately 288K) need perioperative management each year and approximately 1 in 3 (approximately 96K) are considered high-risk patients who need a high-bleed-risk surgery or neuraxial procedure. Perioperative DOAC management is of interest to a wide array of clinicians, including medical, surgical and anesthesia specialties, nurse practitioners, and pharmacists. In support of this statement, the Up-to-Date chapter on Perioperative Anticoagulation is in the top 0.6% (126th of 20,425) of all viewed chapters. However, guidelines provide weak recommendations on perioperative DOAC management in high-bleed-risk patients due to a lack of high-quality data.

There are two competing strategies for DOAC-treated patients who need a high-bleed-risk surgery/neuraxial:

1. PAUSE management is simple and easy to apply as patients having a high-bleed-risk surgery/neuraxial procedure interrupt DOACs for 2 days before and 2 days after surgery without heparin bridging or DOAC level testing. This approach is based on the Perioperative Anticoagulant Use for Surgery Evaluation (PAUSE) study of 3,007-patients with atrial fibrillation (AF) who had elective surgery/procedure.
2. ASRA management is more complex, requiring 72-120 hours DOAC interruption and, in selected patients, pre-operative heparin bridging and DOAC level testing. This management is based on recommendations from the American Society of Regional Anesthesia (ASRA) Guidelines, developed in 2015 and updated in 2018. ASRA's approach is very cautious so as to ensure no residual DOAC level at the time of a high-bleed-risk surgery/neuraxial procedure, using longer pre-operative DOAC interruption intervals.

Clinicians are divided on whether to use PAUSE or ASRA management for perioperative DOAC management in high-bleed-risk patients: Anesthetists strongly favor ASRA, as they consider it safer, in accordance with anesthesia society guidelines, and more prudent medico-legally than PAUSE. On the other hand, internists strongly favor PAUSE, which they consider more evidence-based than ASRA.

As shown in the table below, ASRA management is more complex (variable DOAC interruption) and harder to implement (DOAC testing, heparin bridging) than PAUSE (standard DOAC interruption, no DOAC testing/bridging). Though well-intentioned, ASRA management may not optimize patient safety and, indeed, may hinder adoption of standardized perioperative DOAC management.

ELIGIBILITY:
Inclusion Criteria:

* Adults, age 18 years of age or greater, with AF/flutter (permanent, persistent or paroxysmal) or VTE (leg deep vein thrombosis or pulmonary embolism) that require a full (therapeutic)-dose DOAC regimen, appropriate for age and renal function, comprising one of (a) apixaban 2.5 mg or 5 mg bid; (b) dabigatran 110 mg or 150 mg bid; (c) edoxaban 30 mg or 60 mg daily; or (d) rivaroxaban 15 mg or 20 mg daily
* High-risk patient having an elective high-bleed-risk surgery or any elective surgery with neuraxial anesthesia (epidural, spinal, regional) or any deep nerve root block.

Exclusion Criteria:

* Indication for anticoagulation is unusual site thrombosis (e.g. splanchnic, cerebral, sinus, arm)
* Receiving a low-dose DOAC regimen used for secondary VTE prevention (e.g. rivaroxaban 10 mg daily, apixaban 2.5 mg bid) or another low-dose DOAC regimen (e.g. rivaroxaban 2.5 mg bid)
* CrCL<25mL/min (if on apixaban, edoxaban, rivaroxaban) or <30 mL/min (if on dabigatran)
* cognitive impairment or psychiatric illness that precludes reliable contact during follow up.
* Unable or unwilling to provide consent
* Previous participation in PAUSE 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 920 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients randomized to each study arm with a residual pre-operative DOAC level < 30 ng/mL | Day 1
  The primary outcome in PAUSE-2 will be the proportion of patients with a residual pre-operative DOAC level < 30 ng/mL. Pre-operative DOAC levels will be measured using calibrated anti-Xa assays for direct factor Xa inhibitors (apixaban, edoxaban, rivaroxaban) and will be measured using a dilute thrombin time assay for dabigatran-treated patients.

SECONDARY OUTCOMES:
Proportion of patients with a residual pre-operative DOAC level < 50 ng/mL. | Day 1
  Pre-operative DOAC levels will be measured using calibrated anti-Xa assays for direct factor Xa inhibitors (apixaban, edoxaban, rivaroxaban) and will be measured using a dilute thrombin time assay for dabigatran-treated patients.
Clinically relevant nonmajor bleeding | Day 28
  Any overt bleeding not satisfying the criteria for major bleeding but considered clinically important with one or more of the following criteria met: - Requires minimal medical intervention (blood in urine or stool that is ongoing and requires a sigmoidoscopy, cystoscopy, CBI etc.) by a healthcare professional - Lead to hospitalization or increased level of care - Prompted a face-to-face (ie. not telephone, electronic) evaluation by a physician (this does not include visits prompted by pain, infection, other symptoms etc.)
Arterial thromboembolic Events (ATE) | Day 28
  Any of the following: stroke, systemic embolism, and/or transient ischemic attack. - Ischemic stroke: any new focal neurologic deficit that persists for >24 hours or any new focal neurologic deficit of any duration, that occurs with evidence of acute infarction on computed tomography (CT) or magnetic resonance imaging (MRI) of the brain. - Systemic embolism: symptomatic embolism to upper or lower extremity or abdominal organ, confirmed intra-operatively or by objective imaging (e.g., CT angiography). - Transient ischemic attack: symptomatic focal neurologic deficit (lasting typically <1 hour), that occurs with no evidence of acute infarction on CT/MRI of brain.
Major bleeding | Day 28
  ≥1 of the criteria below: - bleeding that is fatal or is symptomatic and retroperitoneal, intracranial, intraspinal, intraocular, pericardial, intramuscular with compartment syndrome, or intra-articular - non-surgical bleeding causing a drop in hemoglobin ≥20 g/L (1.24 mmol/L) or leading to transfusion ≥2 units whole blood or red cells within 48 hours of the bleed - surgical bleed that leads to intervention (e.g., re-operation) or has one of: (i) interferes with mobilization; (ii) leads to delayed wound healing; or (iii) leads to deep wound infection - surgical site bleeding that is unexpected and prolonged and/or sufficiently large to cause hemodynamic instability associated with: (i) drop in hemoglobin ≥20 g/L (1.24 mmol/L); or (ii) transfusion of ≥2 units whole blood or red cells within 48 hours of the bleed.
Minor bleeding | Day 28
  Any overt bleeding not satisfying the criteria for major and clinically relevant non-major bleeding.
Venous thromboembolic Events (VTE) | Day 28
  Any of the following: symptomatic deep vein thrombosis and/or pulmonary embolism, confirmed by objective imaging studies (e.g., ultrasound, CT pulmonary angiogram).
Myocardial infarction | Day 28
All-cause death | Day 28
  Death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: James Douketis, MD, Principal Investigator — McMaster University/St. Joseph's Healthcare; Joseph Shaw, MD, Principal Investigator — The Ottawa Hospital
Locations (14):
- United States (6):
  - Hartford Health Care, Hartford, Connecticut
  - North Shore University Health, Evanston, Illinois
  - Brigham and Woman's Hospital, Boston, Massachusetts
  - Henry Ford Health Care, Detroit, Michigan
  - Northwell Health System, New York, New York
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
- University of Leuven, Leuven, Belgium, Belgium
- Canada (6):
  - Winnipeg Health Sciences Center, Winnipeg, Manitoba
  - St. Joesph's Healthcare, Hamilton, Ontario
  - Juravinski, Hamilton, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - L'Hospital Montfort, Ottawa, Ontario
  - Toronto General Hospital, Toronto, Ontario
- University of Thessaly, Larissa, Greece, Greece

IPD SHARING:
Plan to Share IPD: No
No IPD data will be shared. All data reported as part of the study is aggregate data.

REFERENCES:
- [Background] Shaw JR, Unachukwu U, Cyr J, Siegal DM, Castellucci LA, Dreden PV, Dowlatshahi D, Buyukdere H, Ramsay T, Carrier M. Effect of PCC on Thrombin Generation among Patients on Factor Xa Inhibitors with Major Bleeding or Needing Urgent Surgery (GAUGE): Design and Rationale. TH Open. 2023 Jul 25;7(3):e229-e240. doi: 10.1055/s-0043-1771300. eCollection 2023 Jul. PMID 37497426
- [Background] Shaw JR, Castellucci LA, Siegal D, Carrier M. DOAC-associated bleeding, hemostatic strategies, and thrombin generation assays - a review of the literature. J Thromb Haemost. 2023 Mar;21(3):433-452. doi: 10.1016/j.jtha.2022.11.029. Epub 2022 Dec 22. PMID 36696204
- [Background] Harenberg J, Beyer-Westendorf J, Crowther M, Douxfils J, Elalamy I, Verhamme P, Bauersachs R, Hetjens S, Weiss C; Working Group Members. Accuracy of a Rapid Diagnostic Test for the Presence of Direct Oral Factor Xa or Thrombin Inhibitors in Urine-A Multicenter Trial. Thromb Haemost. 2020 Jan;120(1):132-140. doi: 10.1055/s-0039-1700545. Epub 2019 Nov 8. PMID 31705521
- [Background] Kim PY, Di Giuseppantonio LR, Wu C, Douketis JD, Gross PL. An assay to measure levels of factor Xa inhibitors in blood and plasma. J Thromb Haemost. 2019 Jul;17(7):1153-1159. doi: 10.1111/jth.14451. Epub 2019 May 10. PMID 30985986
- [Background] Mitrovic D, van Elp M, Veeger N, Lameijer H, Meijer K, van Roon E. Protocols for perioperative management of direct oral anticoagulants in hospitals: opportunities for improvement. Curr Med Res Opin. 2023 Jan;39(1):13-18. doi: 10.1080/03007995.2022.2141962. Epub 2022 Nov 12. PMID 36305802
- [Background] Flaker GC, Theriot P, Binder LG, Dobesh PP, Cuker A, Doherty JU. Management of Periprocedural Anticoagulation: A Survey of Contemporary Practice. J Am Coll Cardiol. 2016 Jul 12;68(2):217-26. doi: 10.1016/j.jacc.2016.04.042. PMID 27386777
- [Background] Kurlander JE, Barnes GD, Anderson MA, Haymart B, Kline-Rogers E, Kaatz S, Saini SD, Krein SL, Richardson CR, Froehlich JB. Mind the gap: results of a multispecialty survey on coordination of care for peri-procedural anticoagulation. J Thromb Thrombolysis. 2018 Apr;45(3):403-409. doi: 10.1007/s11239-018-1625-2. PMID 29423559
- [Background] Wamala H, Scott IA, Caney X. Perioperative management of new oral anticoagulants in patients undergoing elective surgery at a tertiary hospital. Intern Med J. 2017 Dec;47(12):1412-1421. doi: 10.1111/imj.13513. PMID 28589690
- [Background] Korenke M, Samba S, Stam B, Leis A, Kheterpal S, Colquhoun DA. The perioperative management of direct oral anticoagulants, a single center observational study. J Clin Anesth. 2020 Mar;60:92-93. doi: 10.1016/j.jclinane.2019.08.035. Epub 2019 Sep 11. No abstract available. PMID 31520860
- [Background] Nascimento T, Birnie DH, Healey JS, Verma A, Joza J, Bernier ML, Essebag V. Managing novel oral anticoagulants in patients with atrial fibrillation undergoing device surgery: Canadian survey. Can J Cardiol. 2014 Feb;30(2):231-6. doi: 10.1016/j.cjca.2013.11.027. Epub 2013 Dec 4. PMID 24461924
- [Background] Skeith L, Lazo-Langner A, Kovacs MJ. The equipoise of perioperative anticoagulation management: a Canadian cross-sectional survey. J Thromb Thrombolysis. 2014 May;37(4):411-3. doi: 10.1007/s11239-013-0960-6. No abstract available. PMID 23868474
- [Background] Faraoni D, Samama CM, Ranucci M, Dietrich W, Levy JH. Perioperative management of patients receiving new oral anticoagulants: an international survey. Clin Lab Med. 2014 Sep;34(3):637-54. doi: 10.1016/j.cll.2014.06.006. Epub 2014 Jul 23. PMID 25168948
- [Background] Chiang YZ, Al-Niaimi F, Craythorne E, Mallipeddi R. Perioperative management of novel oral anticoagulants in skin surgery: a national survey. Br J Dermatol. 2016 Sep;175(3):615-8. doi: 10.1111/bjd.14462. Epub 2016 Jun 2. No abstract available. PMID 26854272
- [Background] Douketis JD, Spyropoulos AC, Anderson JM, Arnold DM, Bates SM, Blostein M, Carrier M, Caprini JA, Clark NP, Coppens M, Dentali F, Duncan J, Gross PL, Kassis J, Kowalski S, Lee AY, Le Gal G, Le Templier G, Li N, MacKay E, Shah V, Shivakumar S, Solymoss S, Spencer FA, Syed S, Tafur AJ, Vanassche T, Thiele T, Wu C, Yeo E, Schulman S. The Perioperative Anticoagulant Use for Surgery Evaluation (PAUSE) Study for Patients on a Direct Oral Anticoagulant Who Need an Elective Surgery or Procedure: Design and Rationale. Thromb Haemost. 2017 Dec;117(12):2415-2424. doi: 10.1160/TH17-08-0553. Epub 2017 Dec 6. PMID 29212129
- [Background] Merrelaar AE, Bogl MS, Buchtele N, Merrelaar M, Herkner H, Schoergenhofer C, Harenberg J, Douxfils J, Siriez R, Jilma B, Spiel AO, Schwameis M. Performance of a Qualitative Point-of-Care Strip Test to Detect DOAC Exposure at the Emergency Department: A Cohort-Type Cross-Sectional Diagnostic Accuracy Study. Thromb Haemost. 2022 Oct;122(10):1723-1731. doi: 10.1055/s-0042-1750327. Epub 2022 Jul 4. PMID 35785816
- [Background] Lessire S, Douxfils J, Dincq AS, Mullier F. Periprocedural Management of Direct Oral Anticoagulants Should Be Guided by Accurate Laboratory Tests. Reg Anesth Pain Med. 2016 Nov/Dec;41(6):787-788. doi: 10.1097/AAP.0000000000000448. No abstract available. PMID 27662062
- [Background] Douxfils J, Adcock DM, Bates SM, Favaloro EJ, Gouin-Thibault I, Guillermo C, Kawai Y, Lindhoff-Last E, Kitchen S, Gosselin RC. 2021 Update of the International Council for Standardization in Haematology Recommendations for Laboratory Measurement of Direct Oral Anticoagulants. Thromb Haemost. 2021 Aug;121(8):1008-1020. doi: 10.1055/a-1450-8178. Epub 2021 May 30. PMID 33742436
- [Background] Cuker A, Burnett A, Triller D, Crowther M, Ansell J, Van Cott EM, Wirth D, Kaatz S. Reversal of direct oral anticoagulants: Guidance from the Anticoagulation Forum. Am J Hematol. 2019 Jun;94(6):697-709. doi: 10.1002/ajh.25475. Epub 2019 Apr 16. PMID 30916798
- [Background] Spyropoulos AC, Giannis D, Cohen J, John S, Myrka A, Inlall D, Qiu M, Akgul S, Hyman RJ, Wang JJ. Implementation of the Management of Anticoagulation in the Periprocedural Period App Into an Electronic Health Record: A Prospective Cohort Study. Clin Appl Thromb Hemost. 2020 Jan-Dec;26:1076029620925910. doi: 10.1177/1076029620925910. PMID 32633538
- [Background] Lee J, Kong X, Haymart B, Kline-Rogers E, Kaatz S, Shah V, Ali MA, Kozlowski J, Froehlich J, Barnes GD. Outcomes in patients undergoing periprocedural interruption of warfarin or direct oral anticoagulants. J Thromb Haemost. 2022 Nov;20(11):2571-2578. doi: 10.1111/jth.15850. Epub 2022 Sep 1. PMID 35962753
- [Background] Douketis JD, Spyropoulos AC, Duncan J, Carrier M, Le Gal G, Tafur AJ, Vanassche T, Verhamme P, Shivakumar S, Gross PL, Lee AYY, Yeo E, Solymoss S, Kassis J, Le Templier G, Kowalski S, Blostein M, Shah V, MacKay E, Wu C, Clark NP, Bates SM, Spencer FA, Arnaoutoglou E, Coppens M, Arnold DM, Caprini JA, Li N, Moffat KA, Syed S, Schulman S. Perioperative Management of Patients With Atrial Fibrillation Receiving a Direct Oral Anticoagulant. JAMA Intern Med. 2019 Nov 1;179(11):1469-1478. doi: 10.1001/jamainternmed.2019.2431. PMID 31380891
- [Background] Steinberg BA, Hellkamp AS, Lokhnygina Y, Halperin JL, Breithardt G, Passman R, Hankey GJ, Patel MR, Becker RC, Singer DE, Hacke W, Berkowitz SD, Nessel CC, Mahaffey KW, Fox KA, Califf RM, Piccini JP; ROCKET AF Steering Committee and Investigators. Use and outcomes of antiarrhythmic therapy in patients with atrial fibrillation receiving oral anticoagulation: results from the ROCKET AF trial. Heart Rhythm. 2014 Jun;11(6):925-32. doi: 10.1016/j.hrthm.2014.03.006. Epub 2014 May 13. PMID 24833235
- [Background] Valentine D GM, Grissinger M. . Valentine D, Gaunt MJ, Grissinger M. Identifying Patient Harm from Direct Oral Anticoagulants. Available from http://patientsafety.pa.gov/ADVISORIES/Pages/201806_DOACs.aspx. 2020
- [Background] Broderick JP, Bonomo JB, Kissela BM, Khoury JC, Moomaw CJ, Alwell K, Woo D, Flaherty ML, Khatri P, Adeoye O, Ferioli S, Kleindorfer DO. Withdrawal of antithrombotic agents and its impact on ischemic stroke occurrence. Stroke. 2011 Sep;42(9):2509-14. doi: 10.1161/STROKEAHA.110.611905. Epub 2011 Jun 30. PMID 21719769
- [Background] Douketis JD, Spyropoulos AC, Kaatz S, Becker RC, Caprini JA, Dunn AS, Garcia DA, Jacobson A, Jaffer AK, Kong DF, Schulman S, Turpie AG, Hasselblad V, Ortel TL; BRIDGE Investigators. Perioperative Bridging Anticoagulation in Patients with Atrial Fibrillation. N Engl J Med. 2015 Aug 27;373(9):823-33. doi: 10.1056/NEJMoa1501035. Epub 2015 Jun 22. PMID 26095867
- [Background] Spyropoulos AC, Al-Badri A, Sherwood MW, Douketis JD. Periprocedural management of patients receiving a vitamin K antagonist or a direct oral anticoagulant requiring an elective procedure or surgery. J Thromb Haemost. 2016 May;14(5):875-85. doi: 10.1111/jth.13305. Epub 2016 Apr 7. PMID 26988871
- [Background] Douketis JD, Syed S, Li N, Narouze S, Radwi M, Duncan J, Schulman S, Spyropoulos AC. A physician survey of perioperative neuraxial anesthesia management in patients on a direct oral anticoagulant. Res Pract Thromb Haemost. 2020 Dec 16;5(1):159-167. doi: 10.1002/rth2.12430. eCollection 2021 Jan. PMID 33537540
- [Background] Albaladejo P, Bonhomme F, Blais N, Collet JP, Faraoni D, Fontana P, Godier A, Llau J, Longrois D, Marret E, Mismetti P, Rosencher N, Roullet S, Samama CM, Schved JF, Sie P, Steib A, Susen S; French Working Group on Perioperative Hemostasis (GIHP). Management of direct oral anticoagulants in patients undergoing elective surgeries and invasive procedures: Updated guidelines from the French Working Group on Perioperative Hemostasis (GIHP) - September 2015. Anaesth Crit Care Pain Med. 2017 Feb;36(1):73-76. doi: 10.1016/j.accpm.2016.09.002. Epub 2016 Sep 20. PMID 27659969
- [Background] Raval AN, Cigarroa JE, Chung MK, Diaz-Sandoval LJ, Diercks D, Piccini JP, Jung HS, Washam JB, Welch BG, Zazulia AR, Collins SP; American Heart Association Clinical Pharmacology Subcommittee of the Acute Cardiac Care and General Cardiology Committee of the Council on Clinical Cardiology; Council on Cardiovascular Disease in the Young; and Council on Quality of Care and Outcomes Research. Management of Patients on Non-Vitamin K Antagonist Oral Anticoagulants in the Acute Care and Periprocedural Setting: A Scientific Statement From the American Heart Association. Circulation. 2017 Mar 7;135(10):e604-e633. doi: 10.1161/CIR.0000000000000477. Epub 2017 Feb 6. PMID 28167634
- [Background] Doherty JU, Gluckman TJ, Hucker WJ, Januzzi JL Jr, Ortel TL, Saxonhouse SJ, Spinler SA. 2017 ACC Expert Consensus Decision Pathway for Periprocedural Management of Anticoagulation in Patients With Nonvalvular Atrial Fibrillation: A Report of the American College of Cardiology Clinical Expert Consensus Document Task Force. J Am Coll Cardiol. 2017 Feb 21;69(7):871-898. doi: 10.1016/j.jacc.2016.11.024. Epub 2017 Jan 9. PMID 28081965
- [Background] Duffett L. Deep Venous Thrombosis. Ann Intern Med. 2022 Sep;175(9):ITC129-ITC144. doi: 10.7326/AITC202209200. Epub 2022 Sep 13. PMID 36095313
- [Background] Heit JA, Spencer FA, White RH. The epidemiology of venous thromboembolism. J Thromb Thrombolysis. 2016 Jan;41(1):3-14. doi: 10.1007/s11239-015-1311-6. PMID 26780736
- [Background] Barnes GD, Lucas E, Alexander GC, Goldberger ZD. National Trends in Ambulatory Oral Anticoagulant Use. Am J Med. 2015 Dec;128(12):1300-5.e2. doi: 10.1016/j.amjmed.2015.05.044. Epub 2015 Jul 2. PMID 26144101
- [Background] Weitz JI, Semchuk W, Turpie AG, Fisher WD, Kong C, Ciaccia A, Cairns JA. Trends in Prescribing Oral Anticoagulants in Canada, 2008-2014. Clin Ther. 2015 Nov 1;37(11):2506-2514.e4. doi: 10.1016/j.clinthera.2015.09.008. Epub 2015 Oct 16. PMID 26481493
- [Background] Gao L, Tadrous M, Knowles S, Mamdani M, Paterson JM, Juurlink D, Gomes T. Prior Authorization and Canadian Public Utilization of Direct-Acting Oral Anticoagulants. Healthc Policy. 2017 Nov;13(2):68-78. doi: 10.12927/hcpol.2017.25321. PMID 29274228
- [Background] Healey JS, Eikelboom J, Douketis J, Wallentin L, Oldgren J, Yang S, Themeles E, Heidbuchel H, Avezum A, Reilly P, Connolly SJ, Yusuf S, Ezekowitz M; RE-LY Investigators. Periprocedural bleeding and thromboembolic events with dabigatran compared with warfarin: results from the Randomized Evaluation of Long-Term Anticoagulation Therapy (RE-LY) randomized trial. Circulation. 2012 Jul 17;126(3):343-8. doi: 10.1161/CIRCULATIONAHA.111.090464. Epub 2012 Jun 14. PMID 22700854
- [Background] Douketis JD, Spyropoulos AC, Spencer FA, Mayr M, Jaffer AK, Eckman MH, Dunn AS, Kunz R. Perioperative management of antithrombotic therapy: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e326S-e350S. doi: 10.1378/chest.11-2298. PMID 22315266
- [Background] Proietti M, Laroche C, Opolski G, Maggioni AP, Boriani G, Lip GYH; AF Gen Pilot Investigators. 'Real-world' atrial fibrillation management in Europe: observations from the 2-year follow-up of the EURObservational Research Programme-Atrial Fibrillation General Registry Pilot Phase. Europace. 2017 May 1;19(5):722-733. doi: 10.1093/europace/euw112. PMID 27194538
- [Background] Steinberg BA, Gao H, Shrader P, Pieper K, Thomas L, Camm AJ, Ezekowitz MD, Fonarow GC, Gersh BJ, Goldhaber S, Haas S, Hacke W, Kowey PR, Ansell J, Mahaffey KW, Naccarelli G, Reiffel JA, Turpie A, Verheugt F, Piccini JP, Kakkar A, Peterson ED, Fox KAA; GARFIELD-AF; ORBIT-AF Investigators. International trends in clinical characteristics and oral anticoagulation treatment for patients with atrial fibrillation: Results from the GARFIELD-AF, ORBIT-AF I, and ORBIT-AF II registries. Am Heart J. 2017 Dec;194:132-140. doi: 10.1016/j.ahj.2017.08.011. Epub 2017 Aug 24. PMID 29223431
- [Background] Williams BA, Honushefsky AM, Berger PB. Temporal Trends in the Incidence, Prevalence, and Survival of Patients With Atrial Fibrillation From 2004 to 2016. Am J Cardiol. 2017 Dec 1;120(11):1961-1965. doi: 10.1016/j.amjcard.2017.08.014. Epub 2017 Aug 30. PMID 29033050
- [Background] Colilla S, Crow A, Petkun W, Singer DE, Simon T, Liu X. Estimates of current and future incidence and prevalence of atrial fibrillation in the U.S. adult population. Am J Cardiol. 2013 Oct 15;112(8):1142-7. doi: 10.1016/j.amjcard.2013.05.063. Epub 2013 Jul 4. PMID 23831166
- [Background] Halvorsen S, Mehilli J, Cassese S, Hall TS, Abdelhamid M, Barbato E, De Hert S, de Laval I, Geisler T, Hinterbuchner L, Ibanez B, Lenarczyk R, Mansmann UR, McGreavy P, Mueller C, Muneretto C, Niessner A, Potpara TS, Ristic A, Sade LE, Schirmer H, Schupke S, Sillesen H, Skulstad H, Torracca L, Tutarel O, Van Der Meer P, Wojakowski W, Zacharowski K; ESC Scientific Document Group. 2022 ESC Guidelines on cardiovascular assessment and management of patients undergoing non-cardiac surgery. Eur Heart J. 2022 Oct 14;43(39):3826-3924. doi: 10.1093/eurheartj/ehac270. No abstract available. PMID 36017553
- [Background] Parks AL, Fang MC. Periprocedural Anticoagulation. Ann Intern Med. 2023 Apr;176(4):ITC49-ITC64. doi: 10.7326/AITC202304180. Epub 2023 Apr 11. PMID 37037035
- [Background] Narouze S, Benzon HT, Provenzano DA, Buvanendran A, De Andres J, Deer TR, Rauck R, Huntoon MA. Interventional spine and pain procedures in patients on antiplatelet and anticoagulant medications: guidelines from the American Society of Regional Anesthesia and Pain Medicine, the European Society of Regional Anaesthesia and Pain Therapy, the American Academy of Pain Medicine, the International Neuromodulation Society, the North American Neuromodulation Society, and the World Institute of Pain. Reg Anesth Pain Med. 2015 May-Jun;40(3):182-212. doi: 10.1097/AAP.0000000000000223. PMID 25899949
- [Background] Narouze S, Benzon HT, Provenzano D, Buvanendran A, De Andres J, Deer T, Rauck R, Huntoon MA. Interventional Spine and Pain Procedures in Patients on Antiplatelet and Anticoagulant Medications (Second Edition): Guidelines From the American Society of Regional Anesthesia and Pain Medicine, the European Society of Regional Anaesthesia and Pain Therapy, the American Academy of Pain Medicine, the International Neuromodulation Society, the North American Neuromodulation Society, and the World Institute of Pain. Reg Anesth Pain Med. 2018 Apr;43(3):225-262. doi: 10.1097/AAP.0000000000000700. PMID 29278603
- [Background] Douketis JD, Spyropoulos AC, Murad MH, Arcelus JI, Dager WE, Dunn AS, Fargo RA, Levy JH, Samama CM, Shah SH, Sherwood MW, Tafur AJ, Tang LV, Moores LK. Perioperative Management of Antithrombotic Therapy: An American College of Chest Physicians Clinical Practice Guideline. Chest. 2022 Nov;162(5):e207-e243. doi: 10.1016/j.chest.2022.07.025. Epub 2022 Aug 11. PMID 35964704